CLINICAL TRIAL: NCT01463462
Title: Use of the Electronic Catheter Stethoscope for the Detection of Urinary Tract Injury During Gynecologic Surgery
Brief Title: Electronic Catheter Stethoscope
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: USF IRB 00001841
Record Dates: First submitted 2011-10-19; First posted 2011-11-02 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Pelvic Organ Prolapse; Gynecologic Cancers; Uterine Leiomyomata; Adenomyosis; Endometrial Hyperplasia; Other Abnormal Uterine and Vaginal Bleeding; Pelvic Mass; Pelvic Pain
MeSH Terms: conditions — Pelvic Organ Prolapse; Myofibroma; Adenomyosis; Endometrial Hyperplasia; Uterine Hemorrhage; Pelvic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Electronic Catheter Stethoscope

SUMMARY:
This is an observational, exploratory study designed to collect (record) and analyze normal and abnormal sound data from the human bladder during surgery using a novel sensor-based catheter system (Electronic Catheter Stethoscope) and to develop algorithms to detect changes of baseline bladder and ureteral function. The Electronic Catheter Stethoscope device will measure acoustic and pressure data within the bladder. The measurements will be used to detect any leakage from the bladder and/or changes in baseline ureteral flow by correlation of sound data with surgical data reported by the surgeon. These data will be used to develop algorithms to detect changes of baseline bladder and ureteral function. The algorithms will be tested in future clinical trials.

ELIGIBILITY:
Inclusion Criteria

* age 18 or older
* plan to have one of the following types of surgery:

  * laparoscopic or abdominal gynecological surgery
  * vaginal surgery
* able to provide written informed consent

Exclusion Criteria

* under 18 years of age
* bilateral tubal ligation as the single reason for surgery
* current pregnancy
* unable to provide written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current patients having gynecological surgery
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
bladder and ureter sounds during pelvic surgery. | from time of bladder catheter placement and initiation of recording during surgery to completion of pelvic surgery (within 8 hours)

SECONDARY OUTCOMES:
changes from baseline bladder and ureteral function sounds | from time of bladder catheter placement and initiation of recording during surgery to completion of pelvic surgery (within 8 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Hart, MD, Principal Investigator — University of South Florida
Locations (1):
- Women's Center Operating Rooms at the Tampa General Hospital, Tampa, Florida, United States